CLINICAL TRIAL: NCT02351804
Title: Does Perineural Dexamethasone Prolong Duration of an Adductor Canal Block When Controlling for a Systemic Effect? A Paired, Randomized, Blinded, Study in Healthy Volunteers
Brief Title: Does Perineural Dexamethasone Prolong Duration of a Nerve Block?
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Pia Jaeger, Coordinating Investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SM2-PJ-14; 2014-004879-23 (EudraCT Number)
Record Dates: First submitted 2015-01-27; First posted 2015-01-30 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Healthy Volunteers
Keywords: US-guided peripheral nerve block; Anesthetics, Local; duration; Sensation; adductor canal block; lower limb; Adjuvants, Anesthesia
MeSH Terms: interventions — Ropivacaine; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ropivacaine + dexamethasone (Experimental): 20 ml ropivacaine 0.5% + 0.5 ml dexamethasone 4 mg7ml
  Interventions: Drug: Ropivacaine + dexamethasone
- Ropivacaine + placebo (Placebo Comparator): 20 ml ropivacaine 0.5% + 0.5 ml isotonic saline ad
  Interventions: Drug: Ropivacaine + placebo

INTERVENTIONS:
Drug: Ropivacaine + dexamethasone — Adductor canal block, single bolus
  Arms: Ropivacaine + dexamethasone
Drug: Ropivacaine + placebo — Adductor canal block, single bolus
  Arms: Ropivacaine + placebo

SUMMARY:
The purpose of this study is to investigate whether dexamethasone as an adjuvant to ropivacaine for adductor canal block increases duration of the sensory block, when controlling for a systemic effect using a paired design and bilateral blocks.

The investigators hypothesize that adding dexamethasone to ropivacaine will prolong block duration compared with ropivacaine + placebo.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists class 1
* Body Mass Index 18-30

Exclusion Criteria:

* Allergy to study medication
* Earlier trauma or surgery to lower limb
* Diabetes Mellitus
* Alcohol or drug abuse
* Daily intake of opioids or steroids last 4 weeks
* Daily intake of any analgesics last 48 hours

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Difference in duration of sensory block between dexamethasone and placebo assessed as cold sensation with an alcohol swab | 0-36 hours
  Duration is defined as time from block performance until recovery of cold sensation to an alcohol swab, assessed every hour post-block (and every half hour when pain scores during the tonic heat stimulation test is above 0, except at 2 and 3 hours post block where there will be a break and no assessments will be performed.

SECONDARY OUTCOMES:
Difference between dexamethasone and placebo in the duration of a sensory block assessed by pin-prick | 0-36 hours
  Duration is defined as time from block performance until recovery of normal sensation, assessed on the hour post block (except at 2 and 3 hours post block where there will be a break and no assessments will be performed).
Difference between dexamethasone and placebo in the duration of a sensory block assessed as maximum pain during a tonic heat stimulation test | 0-36 hours
  Duration is defined as time from block performance until recovery of normal sensation, assessed on the hour post block (except at 2 and 3 hours post block where there will be a break and no assessments will be performed).
  Recovery of normal sensation is defined as VAS pain scores ± 10 mm of the pre-block value.
Difference between dexamethasone and placebo in the duration of a sensory block assessed as warmth detection threshold | 0-36 hours
  Duration is defined as time from block performance until recovery of normal sensation, assessed on the hour post block (except at 2 and 3 hours post block where there will be a break and no assessments will be performed and only assessed if pain scores during tonic heat stimulation is above 0 ).
  Recovery of normal sensation is defined as detection thresholds of ± 2 degrees C of the pre-block value.
Difference between dexamethasone and placebo in the duration of a sensory block assessed as heat pain detection threshold | 0-36 hours
  Duration is defined as time from block performance until recovery of normal sensation, assessed on the hour post block (except at 2 and 3 hours post block where there will be a break and no assessments will be performed and only assessed if pain scores during tonic heat stimulation is above 0 ).
  Recovery of normal sensation is defined as detection thresholds of ± 2 degrees C of the pre-block value.
Difference in maximum pain scores between dexamethasone and placebo during block and after recovery of normal sensation | 0-36 hours
  Pain scores during a tonic heat stimulation will be compared at 4 h post block and 1 h after pain scores have returned to the pre-block values.

CONTACTS AND LOCATIONS:
Overall Officials: Pia Jæger, MD, PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Department of Anaesthesia-Surgery-Intensive Care, Gentofte Hospital, Gentofte Municipality, Hellerup, Denmark